CLINICAL TRIAL: NCT04829565
Title: Assessment of Pain After Intra-articular Botulinum Toxin Injections in Carpometacarpal Osteoarthritis of the Thumb
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-AOI-11
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Rhizarthrosis
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin (Experimental): 50 IU of botulinum toxin
  Interventions: Drug: Botulinum toxin
- placebo (Placebo Comparator): 50 IU of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin — echo-guided injection into the trapezo-medial-phalangeal jointof 0.5 ml of botulinum toxin 50 IU
  Arms: botulinum toxin
Drug: Placebo — echo-guided injection into the trapezo-medial-phalangeal jointof 0.5 ml of placebo
  Arms: placebo

SUMMARY:
Only 4 randomized controlled clinical trials have been published to date to assess the short-term effectiveness of intra-articular Botulinum Toxin injection on pain, function and quality of life in patients suffering from chronic knee pain related or not to knee osteoarthritis and also in the context of ankle osteoarthritis. The analgesic properties and the reported safety make intra-articular Botulinum toxin a strong candidate in the treatment of symptomatic manifestations of osteoarthritis disease and more particularly in certain locations such as the trapezo-metacarpal joint. Investigators hypothesize that injection of intra-articular Botulinum toxin into the trapezo-metacarpal joint will be of benefit in reducing pain and improving function in patients with rhizarthrosis. Investigators will begin a monocentric randomized controlled trial comparing intra-articular injections of Botulinum toxin and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old
* Patient with rhizarthrosis objectified by interrogation, radiography with at least 2 of the following criteria: osteophyte, joint space narrowing, subchondral sclerosis or geode
* Patient who has had an X-ray of the wrist (face, profile and Kapandji incidence) to estimate the severity of the rhizarthrosis.
* Patient with signed informed consent.
* Visual analog scale (VAS) of pain > 4
* Failure of well-conducted drug treatments with level 1 and 2 analgesics, anti-inflammatory drugs and orthotic devices
* Patients must have stopped all corticosteroid or non-steroidal anti-inflammatory drugs therapy within the last 48 hours.
* Patient affiliated with a Social Security plan
* Patient who can understand the study instructions
* Patient on effective contraception for more than one month according to the marketing authorization (Pill, intrauterine device, vaginal ring, contraceptive skin patch, hormonal subcutaneous implant)
* Infertile patients in connection with surgery (tubal ligation, oophorectomy, adnexectomy, hysterectomy)

Exclusion Criteria:

* History of surgery of the thumb column
* Patient who has received an intra-articular trapezoidal metacarpal injection of corticoids, botulinum toxin or hyaluronic acid or other product within the last 6 months.
* Patient who has received a Botulinum toxin injection at any site within the last 3 months
* Myasthenia or Lambert-Eaton disease, neuromuscular dysfunction, hypersensitivity to incobotulinumtoxin A, severe respiratory disorder or severe swallowing disorder
* Patients with hypersensitivity to botulinum toxin or to any of the excipients (human albumin sucrose)
* Patient with an infection or inflammation at the injection site concerned
* Pregnant or breastfeeding women (a urine pregnancy test will be performed)
* Patients with chronic inflammatory joint disease or microcrystalline pathology
* Current participation or less than 30 days of participation in a clinical drug trial
* Any medical or psychiatric condition that could prevent the proper understanding and conduct of the treatment and study (adult under guardianship)
* Patient who wishes to discontinue contraception during the study
* Patients at high risk of bleeding complications from the intra-articular injection (hemophilia, anticoagulant treatment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale at 3 months | 3 months after the injection
  Evolution of the initial pain by Visual Analogue Scale compared to that measured at 3 months after the injection. Score from 0 to 10. 0 corresponds to the absence of pain and 10 to the maximum imaginable pain.

SECONDARY OUTCOMES:
Dreiser test evaluation | 3 months after the injection
  Dreiser test evaluation (functional index evaluation) at 3 months
adverse events | through study completion, an average of 3 months
  Collecting adverse events
Visual Analogue Scale at 8 weeks | 8 weeks after the injection
  Evaluation of pain by Visual Analogue Scale at 8 weeks. Score from 0 to 10. 0 corresponds to the absence of pain and 10 to the maximum imaginable pain.
intake of analgesic and anti-inflammatory drugs during the study period | from the injection at Month 0 to the evaluation at Month 3, assessed up to 3 months
  Evaluate the intake of analgesic and anti-inflammatory drugs during the study period: collection of the consumption of analgesics and non-steroidal anti-inflammatory drugs in the patient's diary (international non-proprietary name, dosage, date and time) from the injection at Month 0 to the evaluation at Month 3
sleep quality | 3 months after the injection
  sleep quality (Spiegel sleep questionnaire ) at 3 months
quality of life evaluation | 3 months after the injection
  quality of life (SF-36 scale -) at 3 months. a score for each dimension of the SF-36 was calculated, ranging from 0 to 100. A low score reflects a perception of poor health, loss of function, and presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blanc, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, PACA, France